CLINICAL TRIAL: NCT02728414
Title: Probiotics Effect on Glucose and Lipid Metabolism and Gut Microbiota in Patients With Type 2 Diabetes: a Randomized, Double-blind Controlled Trial
Brief Title: Probiotics Effect on Glucose and Lipid Metabolism and Gut Microbiota in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTD01
Record Dates: First submitted 2016-03-25; First posted 2016-04-05 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2, Probiotics, Treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- probiotics (Experimental): the patients in this arm will receive probiotics with a dose for 2g/d for 3 months.
  Interventions: Dietary Supplement: probiotics
- placebo (Other): the patients in this arm will receive placebo with similar appearance of probiotics.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotics — the patients in this arm will receive probiotics with a dose for 2g/d for 3 months.
  Arms: probiotics
Dietary Supplement: placebo — the patients in this arm will receive placebo intervention
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether the probiotics is effective in the treatment of type 2 diabetes.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of probiotics on the improvement of glucose and lipid metabolism, as well as the gut microbiota.Baseline, 1 month and 3 month data will be collected and put into analysis to provide some suggestions on the probiotics use in the clinical practice for type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-80 years
2. Confirmed type 2 diabetes patients with Oral antidiabetic agents
3. Agree to cooperate in the trial
4. Provision of written informed consent

Exclusion Criteria:

1. With chronic gastrointestinal diseases, severe immune deficiency, lactose intolerance
2. Type 1 diabetes
3. Treated with insulin or an insulin analogue in the last 6 months
4. Use antibiotics, bacteriostatic agents (eg berberine), lipid-lowering drugs, antacids, H2 Blockers, proton pump inhibitors, corticosteroids or sex hormones
5. Use any probiotics in the last 3 months
6. Participating in any other clinical trials
7. Was not able to insist until the end
8. Pregnant and lactating women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline in fasting blood-glucose at 1 month | 1 month
  change of the fasting blood-glucose will be calculated at 1 month in comparison with the baseline
change from baseline in fasting blood-glucose at 3 months | 3 months
  change of the fasting blood-glucose will be calculated at 3 months in comparison with the baseline
change from baseline in glycosylated hemoglobin change at 1 month | 1 month
  change of the glycosylated hemoglobin will be calculated at 1 month in comparison with the baseline
change from baseline in glycosylated hemoglobin change at 3 months | 3 months
  change of the glycosylated hemoglobin will be calculated at 3 months in comparison with the baseline

SECONDARY OUTCOMES:
change from baseline in gut microbiota at 1 month | 1 month
  study the microbiota change of stool samples at 1 month in comparison with the baseline
change from baseline in gut microbiota at 3 months | 3 months
  study the microbiota change of stool samples at 3 months in comparison with the baseline
change from baseline in triglyceride at 1 month | 1 month
change from baseline in triglyceride at 3 months | 3 months
change from baseline in cholesterol at 1 month | 1 month
change from baseline in cholesterol at 3 months | 3 months
change from baseline in high-density lipoprotein at 1 month | 1 month
change from baseline in high-density lipoprotein at 3 months | 3 months
change from baseline in low-density lipoprotein at 1 month | 1 month
change from baseline in low-density lipoprotein at 3 months | 3 months
change from baseline in glutamic oxalacetic transaminase at 1 month | 1 month
change from baseline in glutamic oxalacetic transaminase at 3 months | 3 months
change from baseline in alkaline transaminase at 1 month | 1 month
change from baseline in alkaline transaminase at 3 months | 3 months
change from baseline in alkaline phosphatase at 1 month | 1 month
change from baseline in alkaline phosphatase at 3 months | 3 months
change from baseline in superoxide dismutase at 1 month | 1 month
change from baseline in superoxide dismutase at 3 months | 3 months
change from baseline in C-reactive protein at 1 month | 1 month
change from baseline in C-reactive protein at 3 months | 3 months
change from baseline in uric acid at 1 month | 1 month
change from baseline in uric acid at 3 months | 3 months
change from baseline in tumor necrosis factor-a at 1 month | 1 month
change from baseline in tumor necrosis factor-a at 3 months | 3 months
change from baseline in interleukin-6 at 1 month | 1 month
change from baseline in interleukin-6 at 3 months | 3 months
change from baseline in interleukin-8 at 1 month | 1 month
change from baseline in interleukin-8 at 3 months | 3 months
change from baseline in fasting insulin at 1 month | 1 month
change from baseline in fasting insulin at 3 months | 3 months
change from baseline in c peptide at 1 month | 1 month
change from baseline in c peptide at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Huanlong Qin, PhD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided